CLINICAL TRIAL: NCT05961488
Title: Performance of Coronary CT Angiography to Rule Out Coronary Artery Disease After Out-of-hospital Cardiac Arrest
Acronym: PERFECCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PA23075
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Out of Hospital Cardiac Arrest Without ST-segment Elevation
Keywords: Cardiac arrest; Diagnostic accuracy; Coronary computarized tomography angiogram; Coronary Calcium Score; Non-ST Elevated Myocardial Infarction
MeSH Terms: conditions — Heart Arrest; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental)
  Interventions: Other: Coronary Calcium Score and Coronary CT angiogram

INTERVENTIONS:
Other: Coronary Calcium Score and Coronary CT angiogram — Introduction of early Coronary CT angiogram and Coronary Calcium Score in the first days after a resuscitated out-of-hospital cardiac arrest.

SUMMARY:
Out-of-hospital cardiac arrest (OHCA) has multiple etiologies. In the absence of ST-elevation myocardial infarction, percutaneous coronary intervention (PCI) is delayed. This study aims to determine the diagnostic accuracy of Coronary Calcium Score (CCS) and Coronary CT Angiogram (CCTA) to rule out a coronary artery disease (CAD) in the first days after an OHCA.

DETAILED DESCRIPTION:
Each year, 50.000 out-of-hospital cardiac arrest (OHCA) occur in France. Acute myocardial infarction (AMI) is one of the most frequent etiology of OHCA. When a cardiac arrest is due to a ST-elevation myocardial infarction (STEMI), a percutaneous coronary intervention (PCI) is realized in emergency. However, without ST-elevation, PCI timing is unclear. 2020 European Society Recommandations suggest that PCI should not be realized in emergency, based on Lemkes and al. clinical trial. But there is scarce evidence about the exact timing to realize PCI. Electrocardiogram, troponin level, and echocardiography are unprecise to rule-out an ischemic etiology of cardiac arrest.

A brain CT-scan and a CT-pulmonary angiogram are recommended in first place, to identify the etiology of the cardiac arrest if there is no ST-elevation nor obvious causes. Nevertheless, in the absence of scanographic abnormality, a differed coronary angiogram should be realized.

We suggest that coronary CT angiogram (CCTA) and coronary calcium score (CCS) are feasible in the first days of hospitalization, and could rule-out a coronary artery disease (CAD). The aim of the study is to avoid an invasive coronary exploration, and to have a quick answer about anti-thrombotic treatments management.

ELIGIBILITY:
Inclusion criteria :

* Patients hospitalized in intensive care unit after a resuscitated out-of-hospital cardiac arrest
* No obvious cause for sudden death on anamnestic information, CT brain and CT pulmonary angiogram.
* Absence of ST elevation myocardial infarction

Non-inclusion criteria :

* In-hospital cardiac arrest
* Refractory cardiac arrest
* Indication of immediate coronary angiography
* ST-elevation myocardial infarction or unknown left bundle branch block
* Dynamic or presumably new contiguous ST/T-segment changes
* Cardiogenic shock
* Life-threatening arrhythmias
* Coronary artery bypass graft
* Pregnancy
* Multiple organ failure syndrome
* Know severe chronic kidney disease (GFR <30mL/min/1,73m²)

Exclusion criteria :

* During the Coronary computerized tomographic angiogram :
* Haemodynamic instability requiring high dose of vasopressors (>1µg/kg/min of Norepinephrine)
* Non sinusal cardiac rhythm
* KDIGO 1 Acute kidney injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of Coronary Computerized Tomographic Angiogram to rule-out a coronary stenosis > 50% | During hospitalization (maximum 7 days from ICU admission)

SECONDARY OUTCOMES:
Diagnostic accuracy of Coronary Computerized Tomographic Angiogram to rule-out a coronary stenosis > 70% | During hospitalization (maximum 7 days from ICU admission)
Cororany calcium score associated with coronary stenosis between 50% and 70% | During hospitalization (maximum 7 days from ICU admission)
Diagnostic accuracy of Coronary Computerized Tomographic Angiogram associated with Coronary Calcium Score compared to CCTA performance alone | During hospitalization (maximum 7 days from ICU admission)
Incidence of contrast associated acute kidney injury | Day 15
Comparison of contrast volume between CCTA and percutaneous coronary intervention | During hospitalization (maximum 7 days from ICU admission)
Comparison of radiation dose between CCTA and percutaneous coronary intervention | During hospitalization (maximum 7 days from ICU admission)

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France